CLINICAL TRIAL: NCT02474563
Title: A Prospective, Open-label, Multicenter, Observational Study to Evaluate the Efficacy and Safety of Bortezomib, Melphalan, Prednisone(VMP) for Initial Treatment in Patients With Multiple Myeloma Who do Not Undergo Autologous Stem Cell Transplantation
Brief Title: Observational Study to Evaluate the Efficacy and Safety of Bortezomib, Melphalan, Prednisone (VMP) in Participants With Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR018445; 26866138MMY4056 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2015-06-15; First posted 2015-06-17 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bortezomib; Melphalan; Prednisone
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Melphalan; Prednisone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bortezomib, Melphalan, Prednisone (VMP) Group: Participants will not receive any intervention in this study. Participants receiving VMP therapy for MM that was not eligible for autologous stem cell transplantation will be enrolled in the study.
  Interventions: Drug: Bortezomib; Drug: Melphalan; Drug: Prednisone

INTERVENTIONS:
Drug: Bortezomib — Participants receiving Bortezomib 1.3 milligram per square meter (mg/m2) will be observed in this study.
Drug: Melphalan — Participants receiving Melphalan 9 mg/m^2 will be observed in this study.
Drug: Prednisone — Participants receiving Prednisone 60 mg/m^2 will be observed in this study.

SUMMARY:
The purpose of this study is to assess the 2-year progression-free survival rate.

DETAILED DESCRIPTION:
This was a prospective, open-label, multicenter, observational study. Participants who received bortezomib, Melphalan, Prednisone(VMP) therapy for Multiple myeloma (MM) that was not eligible for autologous stem cell transplantation will be enrolled in the study. The study will consist of Screening phase; VMP therapy phase (9cycles); Follow-up phase (2 years from the day when the first cycle was started). Participants visited each institution for evaluation for 2 years from the date of baseline evaluation and first VMP administration (duration of treatment, 9 cycles; follow-up visits, every 3 months after the end of the treatment). Participants receiving VMP therapy will be primarily evaluated for 2-year progression-free survival rate. Participants safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are naïve to chemotherapy for multiple myeloma and not eligible for autologous stem cell transplantation
* Participants with symptomatic multiple myeloma: a) Intramedullary monoclonal plasma cells greater than or equal to (>=) 10% or histologically confirmed plasmacytoma; b) Presence of monoclonal protein in the serum or urine; c) Myeloma-related organ impairment as defined in protocol
* Participants with presence of an illness that is detectable by definitions as defined in protocol
* Postmenopausal, sterilized or sexually inactive women, including women of childbearing potential who exercise effective contraceptive measures before and during the clinical trial

Exclusion Criteria:

* Participants with previous experience of receiving a therapy for multiple myeloma (excluding radiotherapy and dexamethasone < 160mg in total)
* Participants with severe peripheral neuropathy (Grade >= 2 by NCI CTC version 4.0)
* Pregnant or breastfeeding mothers
* Participants with mental illness that can interfere with his/her cooperation with the therapy or the monitoring conditions of the clinical trial
* Participants with other serious medical conditions (such as uncontrolled hypertension, diabetes mellitus and active infections)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants receiving VMP therapy for MM that was not eligible for autologous stem cell transplantation will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
2-year Progression-free Survival Rate | Up to 2 years
  Progression-free survival rate: the length of time from the day when Bortezomib was first administered to disease progression or death, whichever comes first, in 2 years.

SECONDARY OUTCOMES:
Time to Response | up to 2 years
  Time from the first day of Bortezomib administration to the day of confirmed first response in participants with confirmed response, or to the day of loss to follow-up, disease progression, death or completion of study therapy in participants without response.
Overall Response Rate | up to 2 years
  Percentage of participants who achieved CR, VGPR or PR in 2 years.
Complete Response Rate | up to 2 years
  Percentage of participants who achieved CR as best response.
Time to Next therapy | up to 2 years
  The next therapy after the end of the study therapy was investigated, and the time from the day when the first therapy was started to the day when the next therapy was started was calculated.
Time to Disease Progression | up to 2 years
  Time from the first day of Bortezomib administration to the day of disease progression or relapse from complete response, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (18):
- South Korea (18):
  - Anyang
  - Busan
  - Cheonan
  - Chungcheongbuk-Do
  - Daegu
  - Daejeon
  - Gyeonggi-do
  - Hwasun Gun
  - Iksan
  - Incheon
  - Jeonju
  - Jinju
  - Pucheon
  - Pusan
  - Seongnam
  - Seoul
  - Suwon
  - Ulsan